#### **Informed Consent Form**

## **Study Title:**

A Multilevel Study on the Effects of a Mindfulness-Based Intervention Targeting Psychological Capital on Job Burnout Among Nurses: A Randomized Controlled Trial

Principal Investigator: Dr. Mengjie Xia

Institution: Taizhou University, School of Nursing

Contact Information: xiamengjie@tzc.edu.cn

Date: May 1, 2024

#### Introduction

You are invited to participate in a research study that aims to evaluate the effectiveness of a mindfulness-based intervention in reducing job burnout and improving psychological well-being among nurses. This form provides information about the study, what is involved if you choose to participate, and your rights as a participant.

Please read this form carefully and feel free to ask questions before you decide whether to participate.

# **Purpose of the Study**

The goal of this study is to examine whether daily mindfulness practice can help reduce job burnout and improve psychological capital (such as optimism, resilience, and confidence) in nurses. The study also explores how support from family and leadership may influence nurses' emotional health.

## **Procedures**

If you agree to participate, you will be randomly assigned to one of two groups:

Mindfulness Intervention Group: You will receive access to a mobile app providing guided mindfulness practices (e.g., breathing exercises, body scans, meditation). You will be asked to engage in daily practice for approximately 15–20 minutes over a 40-day period.

Control Group: You will continue your routine clinical duties without any additional training or activities.

## All participants will:

Complete online surveys at 4 time points: before the intervention, end of the intervention (Day 40), and at 2 and 4 months after the intervention.

Be asked to answer questionnaires assessing your mental well-being, burnout level, and mindfulness.

Spend about 10 minutes per survey.

#### **Duration**

Your total participation will last approximately 6 months, including the 40-day intervention period and follow-up assessments.

## **Risks and Discomforts**

There are minimal risks associated with this study. You may experience emotional discomfort when reflecting on work-related stress or burnout. You are free to skip any question or withdraw at any time without penalty. You may contact the research team or the university psychological services if you experience distress.

## **Benefits**

You may benefit from:

- Reduced feelings of job burnout
- Improved emotional regulation and resilience
- Increased psychological capital
- Contributing to knowledge that may benefit other nurses and healthcare professionals

However, benefits are not guaranteed.

# Confidentiality

All information collected in this study will be kept strictly confidential. Your data will be anonymized using unique ID numbers and stored on secure, password-protected servers. Only the research team will have access to identifiable data.

Results may be published in scientific journals or presented at conferences, but no information that could identify you will be disclosed.

## **Voluntary Participation**

Your participation in this study is completely voluntary. You may refuse to participate or withdraw at any time, for any reason, without any consequences to your job, academic standing, or relationship with the institution.

# Compensation

There is no financial compensation for participation in this study. However, participants who complete all assessments may receive a small token of appreciation (e.g., certificate).

## **Contact Information**

If you have questions about the study or your rights as a participant, please contact:

Dr. Mengjie Xia

Email:xiamengjie@tzc.edu.cn

Phone: 13028939108

If you have questions about your rights as a research participant, you may contact the Institutional Review Board (IRB) of Taizhou central hospital.

# **Consent Statement**

By signing below, you confirm that:

- You have read and understood the information provided above.
- You have had the opportunity to ask questions.
- You voluntarily agree to participate in this study.

| Participant's Name (Printed): | |
|-------------------------------|---|
| Signature: | - |
| Date: | |
| Researcher's Name (Printed): | |
| Signature: | - |
| Date: | |